CLINICAL TRIAL: NCT02031289
Title: Impact of Preoperative Treatment of Anemia and Iron Deficiency in Cardiac Surgery on Outcome.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IFA2012/IDCS
Record Dates: First submitted 2013-12-16; First posted 2014-01-09 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Anemia; Iron Deficiency
Keywords: Anemia; Iron deficiency; Cardiac surgery; Perioperative Care
MeSH Terms: conditions — Anemia; Iron Deficiencies | interventions — Erythropoietin; Epoetin Alfa; ferric carboxymaltose; Leucovorin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Anemia (Active Comparator): Hb < 120 g/L in women, Hb < 130 g/L in men Erythropoietin/Ferric carboxymaltose/Vitamin B12/Folic Acid
  Interventions: Drug: Erythropoietin/Ferric carboxymaltose/Vitamin B12/Folic Acid
- Iron deficiency (Active Comparator): ferritin < 100 µg/l Erythropoietin/Ferric carboxymaltose/Vitamin B12/Folic Acid
  Interventions: Drug: Erythropoietin/Ferric carboxymaltose/Vitamin B12/Folic Acid
- Natural comparison group (No Intervention): Patients without anemia or iron deficiency will be observed and the same postoperative measurements performed

INTERVENTIONS:
Drug: Erythropoietin/Ferric carboxymaltose/Vitamin B12/Folic Acid — Treatment ) will be given the day before the operation (day -1) or a maximum of 2 days prior to the operation (day -2) in iron deficiency patients and a maximum of 3 days prior to the operation in anemic patients (day -3).
  Erythropoietin alpha (Eprex, Janssen-Cilag AG, Baar) 40'000 U sc. Ferric carboxymaltose (Ferinject, Vifor (International) AG, St. Gallen) 1000 mg in 100 ml NaCl over 30 min.
  Vitamin B12 (Vitarubin®-superconc., Streuli Pharma AG, Uznach) 1 mg sc. Folic acid (Acidum folicum, Streuli Pharma AG, Uznach) 5 mg po.
  Other Names: Eprex; Ferinject; Vitarubin®-superconc; Acidum folicum
  Arms: Anemia; Iron deficiency

SUMMARY:
We are performing the above prospective randomized trial in 1'000 patients undergoing cardiac surgery. The study will answer the question of whether preoperative treatment of anemia or iron deficiency indeed improves transfusion needs (primary outcome) and important clinical outcomes (secondary outcome) in a large group of cardiac surgical patients. The list of inclusion and exclusion criteria was deliberately chosen short so that this patient group largely reflects today's clinical practice .

* Trial with medical product

DETAILED DESCRIPTION:
Anemic or iron deficiency patients are randomized into treatment and placebo groups. Treatment (see below) will be given the day before the operation (day -1) or a maximum of 2 days prior to the operation (day -2) in iron deficiency patients and a maximum of 3 days prior to the operation in anemic patients (day -3). The treatment will not be disclosed to the patient or the health care workers treating the patients during and after the operation.

Patients without anemia or iron deficiency will also be observed and the same postoperative measurements performed. They will serve as a natural comparison group.

Treatment:

Erythropoietin alpha (Eprex, Janssen-Cilag AG, Baar) 40'000 U sc. Ferric carboxymaltose (Ferinject, Vifor (International) AG, St. Gallen) 1000 mg in 100 ml sodiumchloride (NaCl) over 30 min.

Vitamin B12 (Vitarubin®-superconc., Streuli Pharma AG, Uznach) 1 mg sc. Folic acid (Acidum folicum, Streuli Pharma AG, Uznach) 5 mg po.

The current transfusion and coagulation guidelines of the University Hospital of Zurich are followed in both groups identically. Postoperatively on the regular ward a Hb transfusion trigger of 80 g/L is applied

ELIGIBILITY:
Inclusion criteria:

* Patients undergoing valve- and/or coronary bypass surgery
* Signed patient informed consent
* Only patients will be enrolled who won't have an emergency surgery on the same day

Exclusion criteria:

* Participation in another clinical trial within the last 4 weeks prior to enrollment
* Addiction or other disease that did not allow the patient to assess the nature, scope and possible consequences of the clinical tial
* Patients who do not sign the consent form or may not fully understand from inadequate knowledge of German.
* Patients who have not reached the age of legal majority
* Pregnant or lactating women
* Jehovah's Witnesses
* Patients with endocarditis
* Existing allergy or intolerance to ferric carboxymaltose or mannitol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1003 (Actual)
Dates: Start 2013-12; Primary Completion 2017-12 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Red blood cell (RBC) units transfused | 7 days

SECONDARY OUTCOMES:
Percentage of patients without any RBC transfusions | 90 days
Combined allogeneic transfusions (RBC, FFP( fresh frozen plasma), platelets) | 90 days
Length of stay in the intensive care unit (ICU) | 90 days
Duration of mechanical ventilation | 90 days
Acute kidney failure | 7 days
  RIFLE I, AKIN 2
Major Adverse Cardiac and Cerebrovascular Events (MACCE) | 90 days
  Myocardial infarction, stroke, death
New atrial fibrillation | 90 days
Infections | 7 days
  Pneumonia, hospital acquired Deep Sternal Wound Infection
  Definition of infection: rise in inflammation markers after the initial postoperative period (acute phase reaction) and requires treatment and/ or prolongs days in hospital and/or microbiological confirmation of infection
Thrombotic and thromboembolic complications (90 days) | 90 days
  clinical symptoms and evidence of thrombosis/ embolism in one of the following imaging methods (ultrasound, CT-scan)
Length of stay (LOS) in the hospital | 90 days
Length of hospital stay (in comparison to median LOS published for relevant Swiss-DRGs) | 90 days
In hospital mortality | 90 days
30 day and 90-day mortality | 90 days
Costs (for blood products and pharmaceutical products related to transfusion and anemia management) | 90 days
  Comparison of costs for study medication versus costs for blood products and products related to transfusion
Perioperative Hb concentrations | 90 days
Calculated RBC and blood loss | 90 days
Comparison of the treatment and placebo groups with the natural comparison group | 90 days
Safety and tolerance of administered study drug and placebo | 90 days
  Comparison of all serious adverse events between study drug group and placebo group

CONTACTS AND LOCATIONS:
Overall Officials: Donat R Spahn, Prof MD, Principal Investigator — University Hospital Zurich, Institute of Anaesthesiology
Locations (1):
- University Hospital Zurich, Institute of Anaesthesiology, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Rossler J, Schoenrath F, Seifert B, Kaserer A, Spahn GH, Falk V, Spahn DR. Iron deficiency is associated with higher mortality in patients undergoing cardiac surgery: a prospective study. Br J Anaesth. 2020 Jan;124(1):25-34. doi: 10.1016/j.bja.2019.09.016. Epub 2019 Oct 24. PMID 31668348
- [Derived] Spahn DR, Schoenrath F, Spahn GH, Seifert B, Stein P, Theusinger OM, Kaserer A, Hegemann I, Hofmann A, Maisano F, Falk V. Effect of ultra-short-term treatment of patients with iron deficiency or anaemia undergoing cardiac surgery: a prospective randomised trial. Lancet. 2019 Jun 1;393(10187):2201-2212. doi: 10.1016/S0140-6736(18)32555-8. Epub 2019 Apr 26. PMID 31036337